CLINICAL TRIAL: NCT02679417
Title: The Effects of Type of Exercise on Hepatic Fat Content and Metabolic Profiles in Non-alcoholic Fatty Liver Disease: A Randomized Trial
Brief Title: The Effects of Type of Exercise in Non-alcoholic Fatty Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Phunchai Charatcharoenwitthaya, Principle Investigator, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 183/2558(EC1)
Record Dates: First submitted 2016-01-29; First posted 2016-02-10 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: Aminotransferase; Fibrosis, liver; Anthropometry; Exercise
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- aerobic exercise (Active Comparator): Each participant reach a minimum of 50 minutes of some form of aerobic exercise including running on a treadmill 5 to 7 days per week for 12 weeks under the supervision of fitness center trainers.
  Interventions: Behavioral: exercise
- resistant exercise (Active Comparator): Each participant reach a minimum of 50 minutes of some form of strength training involving repetitions of a resistance training exercise for each major muscle group at an intensity for at least 60% of a one-repetition max, 5 to 7 days per week for 12 weeks under the supervision of fitness center trainers.
  Interventions: Behavioral: exercise

INTERVENTIONS:
Behavioral: exercise — 12 weeks of aerobic or resistant exercise

SUMMARY:
The type of physical activity such as, aerobic or resistant exercise required to reduce liver fat content in patient with non-alcoholic fatty liver disease (NAFLD) remains unclear. The purpose of this study is to determine whether aerobic exercise should provide improvement of hepatic fat content and inflammation as well as metabolic profiles and anthropometric parameters better than resistant exercise.

DETAILED DESCRIPTION:
Increasing prevalence of overweight and obese worldwide, non-alcoholic fatty liver disease (NAFLD) is commonly diagnosed in daily clinical practice. Weight reduction has been the only strategy established thus far to reduce hepatic lipid levels. Thus, dietary restriction and exercise focusing on weight reduction is recommended as the cornerstone for managing NAFLD. Recent reports have indicated that increased exercise greatly reduces hepatic fat accumulation and inflammation and the related oxidative stress levels outweigh those achieved by dietary restriction alone. Clear guidelines for such a "lifestyle physical activity" for NAFLD management are currently lacking. The type of physical activity such as, aerobic or resistant exercise required to reduce liver fat content remains unclear.The purpose of this study is to determine whether aerobic exercise should provide improvement of hepatic fat content and inflammation as well as metabolic profiles and anthropometric parameters better than resistant exercise.

ELIGIBILITY:
Inclusion Criteria:

* Siriraj medical personals
* Ultrasonography show liver steatosis by using ultrasound criteria
* Transient elastography by using the controlled attenuation parameter show moderate degree of fatty accumulation in the liver
* History of alcohol consumption in male <20 g/d, female <10 g/d

Exclusion Criteria:

* Liver disease of other etiology
* Medications that caused fatty accumulation in the liver
* Treated with vitamin E or antidiabetic agents
* Cardiopulmonary diseases or orthopedic conditions that are contraindicated for exercise

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2015-08; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Hepatic fat content as assessed by the controlled attenuation parameter. | 12 weeks
  Hepatic fat content will be assessed with the controlled attenuation parameter (CAP) at baseline and the end of 12 weeks. The CAP measures ultrasonic attenuation in the liver at 3.5 MHz using signals acquired by the FibroScan® M probe based on vibration-controlled transient elastography. The final CAP value, which ranges from 100 to 400 decibels per metre (dB/m), is the median of individual measurements.

SECONDARY OUTCOMES:
Hepatic inflammation as assessed by serum levels of aspartate aminotransferase, alanine aminotransferase, ferritin and c-reactive protein. | 12 weeks
  Venous blood samples will be obtained for aspartate aminotransferase, alanine aminotransferase, ferritin and c-reactive protein to evaluate the evidence of hepatic inflammation at baseline, 4 weeks, 8 weeks and 112 weeks.
Liver fibrosis as assessed by vibration-controlled transient elastography. | 12 weeks
  Liver fibrosis will be acquired by the FibroScan® M probe based on vibration-controlled transient elastography at baseline and the end of 12 weeks. Liver stiffness measurement will be performed by a single operator who is blinded to all clinical data of the patients. Ten successful acquisitions will be performed on each patient. The median value is considered representative of the elastic modulus of the liver expressed in kilopascal (kPa).
Metabolic profiles assessed with the measurement of lipid profiles, plasma glucose, insulin and oral glucose tolerance test. | 12 weeks
  Venous blood samples will be obtained after a 12-hour overnight fast for total cholesterol, triglyceride, high density lipoprotein cholesterol, low density lipoprotein cholesterol, plasma glucose, insulin, and oral glucose tolerance test at baseline and the end of 12 weeks.
Anthropometry and bioelectrical impedance assessed by a bioelectrical fat analyzer. | 12 weeks
  All anthropometric measurements will be performed with the subjects wearing light clothes without shoes at baseline, 4 weeks, 8 weeks and 12 weeks. Height will be measured to the nearest 0.01 m using a calibrated wall-mounted stadiometer. Body weight will be determined to the nearest 0.05 kg using a calibrated balance beam scale. Body mass index will be calculated as weight (kg) divided by the height-squared (m2). Body circumferences will be measured with a flexible tape, with the subject in the upright position at the end of a gentle expiration, at the following levels: waist (midway between the lower rib margin and the superior interior iliac spine) and hip (widest circumference over the great trochanters). Bioelectrical impedance analysis will be performed with the use of a bioelectrical fat analyzer at baseline, 4 weeks, 8 weeks and 12 weeks.
Cardiorespiratory fitness as assessed with maximal oxygen uptake under treadmill test. | 12 weeks
  Cardiorespiratory fitness will be assessed by a trained health technician at baseline and the end of 12 weeks. The protocol of treadmill test include a 2-min warm-up, two 3-min exercise stages, and a 2-min cool down period. The protocol goal is to elicit a heart rate that is approximately 75% of the age-predicted maximum (220-age) by the end of the test. Heart rate will be monitored throughout the test, and blood pressure will be measured at the end of each stage. Maximal oxygen uptake (V·O2max) will be estimated using a calculation.

CONTACTS AND LOCATIONS:
Overall Officials: Phunchai Charatcharoenwitthaya, MD, Principal Investigator — Siriraj Hospital
Locations (1):
- Faculty of Medicine Siriraj Hospital, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chalasani N, Younossi Z, Lavine JE, Diehl AM, Brunt EM, Cusi K, Charlton M, Sanyal AJ. The diagnosis and management of non-alcoholic fatty liver disease: practice Guideline by the American Association for the Study of Liver Diseases, American College of Gastroenterology, and the American Gastroenterological Association. Hepatology. 2012 Jun;55(6):2005-23. doi: 10.1002/hep.25762. No abstract available. PMID 22488764
- [Background] Vernon G, Baranova A, Younossi ZM. Systematic review: the epidemiology and natural history of non-alcoholic fatty liver disease and non-alcoholic steatohepatitis in adults. Aliment Pharmacol Ther. 2011 Aug;34(3):274-85. doi: 10.1111/j.1365-2036.2011.04724.x. Epub 2011 May 30. PMID 21623852
- [Background] Beymer C, Kowdley KV, Larson A, Edmonson P, Dellinger EP, Flum DR. Prevalence and predictors of asymptomatic liver disease in patients undergoing gastric bypass surgery. Arch Surg. 2003 Nov;138(11):1240-4. doi: 10.1001/archsurg.138.11.1240. PMID 14609874
- [Background] Leite NC, Salles GF, Araujo AL, Villela-Nogueira CA, Cardoso CR. Prevalence and associated factors of non-alcoholic fatty liver disease in patients with type-2 diabetes mellitus. Liver Int. 2009 Jan;29(1):113-9. doi: 10.1111/j.1478-3231.2008.01718.x. Epub 2008 Apr 1. PMID 18384521
- [Background] Assy N, Kaita K, Mymin D, Levy C, Rosser B, Minuk G. Fatty infiltration of liver in hyperlipidemic patients. Dig Dis Sci. 2000 Oct;45(10):1929-34. doi: 10.1023/a:1005661516165. PMID 11117562
- [Background] Musso G, Gambino R, Cassader M, Pagano G. Meta-analysis: natural history of non-alcoholic fatty liver disease (NAFLD) and diagnostic accuracy of non-invasive tests for liver disease severity. Ann Med. 2011 Dec;43(8):617-49. doi: 10.3109/07853890.2010.518623. Epub 2010 Nov 2. PMID 21039302
- [Background] Hashimoto E, Yatsuji S, Tobari M, Taniai M, Torii N, Tokushige K, Shiratori K. Hepatocellular carcinoma in patients with nonalcoholic steatohepatitis. J Gastroenterol. 2009;44 Suppl 19:89-95. doi: 10.1007/s00535-008-2262-x. Epub 2009 Jan 16. PMID 19148800
- [Background] Promrat K, Kleiner DE, Niemeier HM, Jackvony E, Kearns M, Wands JR, Fava JL, Wing RR. Randomized controlled trial testing the effects of weight loss on nonalcoholic steatohepatitis. Hepatology. 2010 Jan;51(1):121-9. doi: 10.1002/hep.23276. PMID 19827166
- [Background] Sullivan S, Kirk EP, Mittendorfer B, Patterson BW, Klein S. Randomized trial of exercise effect on intrahepatic triglyceride content and lipid kinetics in nonalcoholic fatty liver disease. Hepatology. 2012 Jun;55(6):1738-45. doi: 10.1002/hep.25548. Epub 2012 Apr 25. PMID 22213436
- [Background] Hallsworth K, Fattakhova G, Hollingsworth KG, Thoma C, Moore S, Taylor R, Day CP, Trenell MI. Resistance exercise reduces liver fat and its mediators in non-alcoholic fatty liver disease independent of weight loss. Gut. 2011 Sep;60(9):1278-83. doi: 10.1136/gut.2011.242073. Epub 2011 Jun 27. PMID 21708823
- [Background] Fealy CE, Haus JM, Solomon TP, Pagadala M, Flask CA, McCullough AJ, Kirwan JP. Short-term exercise reduces markers of hepatocyte apoptosis in nonalcoholic fatty liver disease. J Appl Physiol (1985). 2012 Jul;113(1):1-6. doi: 10.1152/japplphysiol.00127.2012. Epub 2012 May 10. PMID 22582214
- [Background] Jin YJ, Kim KM, Hwang S, Lee SG, Ha TY, Song GW, Jung DH, Kim KH, Yu E, Shim JH, Lim YS, Lee HC, Chung YH, Lee Y, Suh DJ. Exercise and diet modification in non-obese non-alcoholic fatty liver disease: analysis of biopsies of living liver donors. J Gastroenterol Hepatol. 2012 Aug;27(8):1341-7. doi: 10.1111/j.1440-1746.2012.07165.x. PMID 22554085
- [Background] Oh S, Tanaka K, Warabi E, Shoda J. Exercise reduces inflammation and oxidative stress in obesity-related liver diseases. Med Sci Sports Exerc. 2013 Dec;45(12):2214-22. doi: 10.1249/MSS.0b013e31829afc33. PMID 23698242
- [Background] Zelber-Sagi S, Buch A, Yeshua H, Vaisman N, Webb M, Harari G, Kis O, Fliss-Isakov N, Izkhakov E, Halpern Z, Santo E, Oren R, Shibolet O. Effect of resistance training on non-alcoholic fatty-liver disease a randomized-clinical trial. World J Gastroenterol. 2014 Apr 21;20(15):4382-92. doi: 10.3748/wjg.v20.i15.4382. PMID 24764677
- [Background] Bacchi E, Negri C, Targher G, Faccioli N, Lanza M, Zoppini G, Zanolin E, Schena F, Bonora E, Moghetti P. Both resistance training and aerobic training reduce hepatic fat content in type 2 diabetic subjects with nonalcoholic fatty liver disease (the RAED2 Randomized Trial). Hepatology. 2013 Oct;58(4):1287-95. doi: 10.1002/hep.26393. Epub 2013 Aug 22. PMID 23504926
- [Derived] Charatcharoenwitthaya P, Kuljiratitikal K, Aksornchanya O, Chaiyasoot K, Bandidniyamanon W, Charatcharoenwitthaya N. Moderate-Intensity Aerobic vs Resistance Exercise and Dietary Modification in Patients With Nonalcoholic Fatty Liver Disease: A Randomized Clinical Trial. Clin Transl Gastroenterol. 2021 Mar;12(3):e00316. doi: 10.14309/ctg.0000000000000316. PMID 33939383